CLINICAL TRIAL: NCT04742062
Title: First in Human Dose Ascending, Randomized, Placebo-Controlled Clinical Trial to Assess Tolerability and Pharmacokinetics of ApTOLL in Healthy Volunteers
Brief Title: First in Human Clinical Trial of ApTOLL in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: aptaTargets S.L. (Industry)
Collaborators: Ministry of Science and Innovation, Spain (Other Government); Anagram (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ApTOLL-FIH-01
Record Dates: First submitted 2021-01-26; First posted 2021-02-05 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2021-01

CONDITIONS: Stroke
Keywords: Healthy volunteers; ApTOLL
MeSH Terms: conditions — Stroke | interventions — TLR4 antagonist ApTOLL

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ApTOLL single dose (Active Comparator): ApTOLL is administered intravenously in a single ascending dose pattern in seven dose levels (0.7mg - 70mg). Levels 1 - 3 include one subject per level and levels 4 - 7 include six subjects per level (1 sentinel + 5 subjects).
  Interventions: Drug: ApTOLL
- Placebo single dose (Placebo Comparator): Placebo is administered intravenously during seven dose levels. Levels 1 - 3 include one subject per level and levels 4 - 7 include two subjects per level (1 sentinel + 1 subject).
  Interventions: Other: Placebo
- ApTOLL multiple dose (Active Comparator): ApTOLL is administered intravenously every eight hours during 24h (21mg). This arm includes six subjects (1 sentinel + 5 subjects).
  Interventions: Drug: ApTOLL
- Placebo multiple dose (Placebo Comparator): Placebo is administered intravenously every eight hours during 24h. This arm includes twosubjects (1 sentinel + 1 subject).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ApTOLL — ApTOLL is a Toll-like receptor 4 (TLR4) antagonist, a receptor that is involved in innate immune responses but also responds to tissue damage, and therefore it is directly involved in a large number of diseases where the inflammatoryy response is involved. ApTOLL has demonstrated specific binding to human TLR4 as well as a TLR4 antagonistic effect, reducing inflammation and improving outcome after different disease models.
  Arms: ApTOLL multiple dose; ApTOLL single dose
Other: Placebo — 100 mL 0.9% Sodium Chloride solution
  Arms: Placebo multiple dose; Placebo single dose

SUMMARY:
This is a Phase I, first-in-human, dose ascending, randomized, placebo-controlled clinical study to assess the tolerability and pharmacokinetics of ApTOLL in healthy volunteers. ApTOLL is an aptamer able to antagonize TLR4 receptor and, therefore, to reduce the inflammatory response.

DETAILED DESCRIPTION:
This Phase I clinical trial is divided in two parts: the first part (part A) is a single dose escalation study and the second (part B) is a multiple dose study. Both are performed in healthy volunteers.

* First part: a single dose, i.v. administration (slow infusion), dose escalation with a maximum of 7 single dose levels, randomized, double-blind, placebo-controlled (saline solution), in healthy subjects.
* Second part: a multiple dose, i.v. administration (slow infusion), randomized, double-blind, placebo-controlled (saline solution), in healthy subjects.

The main objectives of this study are:

1. To evaluate the tolerability and pharmacokinetic characteristics of ApTOLL in healthy volunteers, after single dose administration in fasting conditions, following an ascending dosing scheme.
2. To evaluate the tolerability and pharmacokinetic characteristics of ApTOLL in healthy volunteers, after multiple dose administration in fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects (women without possibility of becoming pregnant) willing and able to give their written consent to participate in the trial.
2. Healthy subjects aged within: 18 to 55 years (limits included).
3. Clinical history and physical examination results within normality.
4. Vital signs and electrocardiogram without clinically significant pathologic abnormalities and with QTc (Corrected QT space) values lower than 450 ms.
5. Body weight between 65 and 85 kg, inclusive.
6. BMI (Body Mass Index) between 19.0 and 30.0 kg/m2.
7. No clinically significant abnormalities in haematology, biochemistry, serology (Ag HBV (Hepatitis B Virus), HCV (Hepatitis C Virus) antibodies, HIV (Human Immunodeficiency Virus) antibodies) and urine tests.

Exclusion Criteria:

1. Any chronic medical condition (such as type 1 diabetes) requiring chronic treatment.
2. Evidence of active infection requiring antibiotic therapy within 14 days prior to screening.
3. Medical history of vasculitis or any autoimmune disease excluding seasonal allergic rhinitis and childhood history of atopic dermatitis.
4. Subject having at screening examination a sitting blood pressure more than or equal to 140/90 mm Hg or lower than or equal to 90/50 mmHg.
5. Subject having at screening examination a pulse more than 100 beats per minute or a body temperature more than 37.7 °C. or a respiratory rate outside the normal range of (14-20 breath per minute).
6. History of any treatment for cancer within the past 2 years, other than basal cell or squamous cell carcinoma of the skin.
7. Clinically significant abnormalities in screening laboratory tests.
8. Any prescription, over-the-counter and herbal medications within 10 days prior to study dosing.
9. Use of an investigational drug within 3 months prior to dosing in this study.
10. Psychiatric history of current or past psychosis, bipolar disorder, clinical depression, or anxiety disorder requiring chronic medication within the past 5 years.
11. Pregnant or breastfeeding women.
12. History of substance abuse, including alcohol.
13. Smokers.
14. History of substance or drug dependence, or positive urine drug screen at screening visit.
15. History of head injury.
16. History of sensitivity to any drug.
17. Having donated blood in the last month before start of the study.
18. Any reason or opinion of the investigator that would prevent the subject from participation in the study.
19. Inability to follow the instructions or an unwillingness to collaborate during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events as assessed by CTCAE v4.0 | From dosing to follow-up (day 15 after dosing)
  Adverse Events that occur during the study
Peak Plasma Concentration | Predose and at different times up to 72 hours post-dose
  Peak Plasma Concentration (Cmax)
Area under the plasma concentration | Predose and at different times up to 72 hours post-dose
  Area under the plasma concentration versus time curve (AUC)

SECONDARY OUTCOMES:
Vital signs | From screening to follow-up (day 15 after dosing)
  Heart Rate
Vital signs | From screening to follow-up (day 15 after dosing)
  Blood Presure
Vital signs | From screening to follow-up (day 15 after dosing)
  Respiratory Rate
Vital signs | From screening to follow-up (day 15 after dosing)
  Body Temperature
Laboratory determinations | From screening to follow-up (day 15 after dosing)
  Number of patients with treatment-related alterations coagulation parameters (Protrombine Time (PT) and activated Partial Tromboplastine Time (aPTT))
Laboratory determinations | From screening to follow-up (day 15 after dosing)
  Number of patients with treatment-related alterations Complement Factors activation determined in blood

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Ochoa, MD, PhD, Principal Investigator — Clinical Trials Unit. Hospital Universitario La Princesa; Macarena Hernández, PhD, Study Director — aptaTargets S.L.
Locations (1):
- Clinical Pharmacology Department. Hospital Universitario de La Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
All the data from this study are going to be published.

REFERENCES:
- [Derived] Duran-Laforet V, Pena-Martinez C, Garcia-Culebras A, Alzamora L, Moro MA, Lizasoain I. Pathophysiological and pharmacological relevance of TLR4 in peripheral immune cells after stroke. Pharmacol Ther. 2021 Dec;228:107933. doi: 10.1016/j.pharmthera.2021.107933. Epub 2021 Jun 24. PMID 34174279
- See also: Biotechnology company specialized in therapeutic aptamers — http://aptatargets.com